CLINICAL TRIAL: NCT00847834
Title: Multi-center Open Label, Non-comparative Observational Study of Irbesartan-Hydrochlorothiazide in the Treatment of Hypertension in Chinese Population
Brief Title: Irbesartan-Hydrochlorothiazide Phase IV Study: Treatment of Hypertension in Chinese Population
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: L_9292
Record Dates: First submitted 2009-02-18; First posted 2009-02-19 (Estimated); Last update posted 2009-09-15 (Estimated); Status verified 2009-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Irbesartan; Hydrochlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 4 weeks of one tablet Irbesartan 150mg / Hydrochlorothiazide 12.5mg followed by:
  * If DBP<85mmHg: 4 weeks of one tablet of Irbesartan 150mg / Hydrochlorothiazide 12.5mg
  * If DBP≥85mmHg: 4 weeks of one tablet of Irbesartan 150mg / Hydrochlorothiazide 12.5mg + one tablet of Irbesartan 150mg
  Interventions: Drug: Irbesartan 150mg / Hydrochlorothiazide 12.5mg; Drug: Irbesartan 150mg
- 2 (Experimental): 2 weeks of one tablet Irbesartan 150mg / Hydrochlorothiazide 12.5mg followed by 2 weeks of one tablet Irbesartan 150mg / Hydrochlorothiazide 12.5mg + one tablet Irbesartan 150mg followed by:
  * If DBP<85mmHg: 4 weeks of of one tablet Irbesartan 150mg / Hydrochlorothiazide 12.5mg + one tablet Irbesartan 150mg
  * If DBP≥85mmHg: 4 weeks of two tablets Irbesartan 150mg / Hydrochlorothiazide 12.5mg
  Interventions: Drug: Irbesartan 150mg / Hydrochlorothiazide 12.5mg; Drug: Irbesartan 150mg

INTERVENTIONS:
Drug: Irbesartan 150mg / Hydrochlorothiazide 12.5mg — Once a day
Drug: Irbesartan 150mg — Once a day

SUMMARY:
To analyse the control rate of irbesartan/hydrochlorothiazide(HCTZ) (COAPROVEL) in the treatment of patients with mild to moderate primary hypertension.

ELIGIBILITY:
Inclusion criteria:

* Systolic blood pressure < 180 mmHg
* 90 mmHg ≤ Diastolic blood pressure < 110 mmHg

Exclusion criteria:

* Pregnancy or lactation. Women of child bearing potential (not post-menopausal) should be using a reliable contraceptive method
* Known or suspected secondary hypertension (e.g., coarctation of aorta, renovascular stenosis, etc.)
* Presence of clinically significant ventricular or supraventricular arrhythmias, or second or third degree atrioventricular block, or sick sinus syndrome
* ALAT[SGPT]>2 times of upper limit，
* ASAT[SGOT]>2 times of upper limit
* Patients with known renal disease
* Serum potassium > normal upper limit
* Uncontroled BD（FBG>10mmol/L or PBG>12.22mmol/L)
* Patients treated with tricyclic antidepressants
* Clinical hematological disease.
* Patients with a history of irbesartan, or hydrochlorothiazide sensitivity defined as irbesartan, or hydrochlorothiazide discontinuation due to medically significant adverse effects.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 968 (Actual)
Dates: Start 2003-12; Primary Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who reach a diastolic blood pressure <85 mmHg | At 2, 4 and 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ji Jing, Study Director — Sanofi
Locations (1):
- Sanofi aventis administrative office, Beijing, China